CLINICAL TRIAL: NCT06097819
Title: Investigation of the Effect of Occupational Therapy-based Rehabilitative Games on Motor Skills, Proprioception and Cognitive Functions in Individuals With Intellectual Disabilities
Brief Title: Therapy-Based Games' Effects on Motor and Cognitive Skills in Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-212
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Intellectual Disability
Keywords: exergame; Intellectual Disability; Video game based therapy
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile app-based game group (Experimental): The mobile app-based game group will receive the Becure mobile game program in addition to occupational therapy interventions and the sensor-based game application. This program will be implemented for 10 minutes a day, 5 days a week, for a duration of 6 weeks.
  Interventions: Other: Mobile app-based game group
- Supervised combined sensor-based game group (Experimental): A supervised combined sensor-based game intervention based on occupational therapy will be applied to this group. For this group, a supervised combined sensor-based game program was designed in addition to 12 sessions of occupational therapy interventions over 6 weeks, with 2 sessions per week and each session averaging 30 minutes
  Interventions: Other: Supervised combined sensor-based game group
- Individualized occupational therapy group (Experimental): Individualized occupational therapy group will receive occupational therapy sessions. During these sessions, activities that involve weight transfer, balance, fine motor skills, neuromuscular function, and cognitive skills will be implemented. Treatment will be administered for 2 days a week over a period of 6 weeks. Each session will last an average of 30 minutes. A total of 12 occupational therapy sessions will be conducted
  Interventions: Other: Individualized occupational therapy group

INTERVENTIONS:
Other: Mobile app-based game group — Mobile app based game therapy+Occupational therapy+Sensor-based game therapy
  Arms: Mobile app-based game group
Other: Supervised combined sensor-based game group — Occupational therapy+Sensor-based game therapy
  Arms: Supervised combined sensor-based game group
Other: Individualized occupational therapy group — Occupational therapy
  Arms: Individualized occupational therapy group

SUMMARY:
Individuals with intellectual disabilities face challenges in areas of attention, motor skills, and awareness. Among the problems they experience are difficulties in focusing, transitioning from one activity to another, performing tasks in sequence in skills such as copying, reading, and writing. Additionally, they tend to form sentences with misarranged words. Generally, they may present with disorganized or weak handwriting. Other reported issues in this population include coordination problems in extremities and balance disturbances. These essential life skills can impede the individual's ability to move safely. With the recent integration of technology into rehabilitation, new intervention and assessment methods have emerged for occupational therapists. Systems like Microsoft Kinect, Nintendo Wii, Xbox, and Leap Motion are being used in these methods. In the literature, Kwok et al. included 73 participants aged between 60-85 in their study. They examined the connection between swinging speeds while standing on both feet on a balance board and the risk of falling. They concluded that the anterior-posterior swing speed measure derived from the Wii Balance Board (WBB) could complement current clinic-based measurements in predicting future falls among community-dwelling older adults. Reviewing the literature, technological rehabilitation applications are observed to be used in various patient groups. However, studies on occupational therapy-based technological rehabilitation interventions in individuals with intellectual disabilities are limited. To our knowledge, there isn't a study evaluating awareness, cognitive, and physical skills in intellectually disabled individuals using Leapmotion, Xbox, Balanceboard sensors, and mobile games. Based on this information, the aim of our study is to investigate the effects of occupational therapy-based rehabilitative games on motor skills, proprioception, and cognitive functions in individuals with intellectual disabilities.

DETAILED DESCRIPTION:
A total of 45 participants will be included in the study. These 45 participants will be divided into three groups, and each participant will receive an intervention twice a week for six weeks following the initial assessment.

Group → Mobile application-based game group Group → Supervised combined sensor-based game group Group → Individualized occupational therapy group Participants will be assessed both before and after the 12-session intervention. Participants' attention and reaction time will be evaluated using MOXO-dCPT, proprioceptive awareness will be assessed using Becure Extremity ROM, neuromuscular function will be measured using the 30-second sit-to-stand test, and fine motor skills will be assessed using the nine-hole peg test.

Inclusion criteria:

* Being aged between 18 and 30.
* Obtaining an IQ score between 40 and 70 based on the psychiatric evaluation.
* Having mild to moderate intellectual disability.
* Being able to participate in the games.

Exclusion criteria:

* Presence of behavioral disorders.
* Inability to cooperate with the application instructions.
* Individuals with visual problems and sensitivity to light.
* Presence of limiting neurological, vascular, and cardiac problems.

Outcome measures:

Joint position sense: Joint position sense evaluation measures proprioceptive awareness. Individuals are asked to actively reposition to a degree shown to them before the measurement begins. The individual's active repositioning angle is then measured again, and the difference between the required angle and the actual angle is compared. The closer these two values are to each other, the better the individual's proprioceptive awareness. In our study, proprioceptive awareness for shoulder abduction and flexion measurements will be assessed using the Becure Extremity Rom.

Evaluation of Neuromuscular Function

The 30-second sit-to-stand test requires participants to sit down and stand up from a chair as many times as possible within a 30-second time frame. The scores are associated with muscle strength and functionality. This test is a rapid, cost-effective, safe, and commonly used clinical assessment for lower extremity function.

Evaluation of Fine Motor Skills

The Nine Hole Peg Test consists of a platform with nine holes spaced 32mm apart and nine pegs. Individuals are instructed to remove all pegs from the holes as quickly as possible, one by one, and then to pick up each peg and place it back into the holes on the platform in the shortest time possible. The platform is positioned toward the hand being tested, while the pegs are placed towards the individual's midline. Only the evaluated hand performs the test, and the non-evaluated hand is allowed to hold the edge of the platform for stability. Scores are based on the time, recorded in seconds, taken to complete the test activity. Evaluation of Attention and Reaction Time

The MOXO-dCPT is a computer-based test anchored on an online platform comprising eight sections. The auditory and visual distractors present in the test simulate environmental conditions individuals encounter in daily life. Each section contains 53 stimuli. Every stimulus is displayed in the center of the computer screen as either a target or non-target. This is followed by an interval of equal duration where no stimuli are shown, referred to as a "gap". Participants are instructed to press the space bar in response to targets and refrain from pressing it for non-targets. This is done while overlooking a series of visual and auditory distractors (e.g., an animation of a barking dog). The sections of the MOXO-dCPT vary in cognitive challenge. Within the eight sections of this test; the 1st and 8th sections include classic distractors, the 2nd and 3rd sections involve visual distractors, the 4th and 5th sections contain auditory distractors, and the 6th and 7th sections feature combinations of both visual and auditory distractors.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30.
* Having an IQ score between 40-70 as determined by psychiatric evaluation.
* Possessing mild to moderate intellectual disability.
* Being able to participate in games.

Exclusion Criteria:

* Presence of behavioral disorders.
* Inability to cooperate with application instructions.
* Individuals with visual problems and sensitivity to light.
* Functional limitations due to neurological, vascular, and cardiac problems.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Joint position sense | 10 minutes
  Individuals are asked to actively reposition to a degree shown to them before the measurement begins. The individual's active repositioning angle is then measured again, and the difference between the required angle and the actual angle is compared. The closer these two values are to each other, the better the individual's proprioceptive awareness. In our study, proprioceptive awareness for shoulder abduction and flexion measurements will be assessed using the Becure Extremity Rom.
Neuromuscular Function | 10 minutes
  The 30-second sit-to-stand test requires participants to sit down and stand up from a chair as many times as possible within a 30-second time frame. The scores are associated with muscle strength and functionality. This test is a rapid, cost-effective, safe, and commonly used clinical assessment for lower extremity function.
Evaluation of Fine Motor Skills | 15 minutes
  The Nine Hole Peg Test consists of a platform with nine holes spaced 32mm apart and nine pegs. Individuals are instructed to remove all pegs from the holes as quickly as possible, one by one, and then to pick up each peg and place it back into the holes on the platform in the shortest time possible. The platform is positioned toward the hand being tested, while the pegs are placed towards the individual's midline. Only the evaluated hand performs the test, and the non-evaluated hand is allowed to hold the edge of the platform for stability. Scores are based on the time, recorded in seconds, taken to complete the test activity.
Attention and Reaction Time | 20 minutes
  MOXO-dCPT
  The MOXO-dCPT is a computer-based test anchored on an online platform comprising eight sections. The auditory and visual distractors present in the test simulate environmental conditions individuals encounter in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, PhD, Principal Investigator — Medipol University
Locations (1):
- Bağcılar Municipality Feyzullah Kıyıklık Palace for the Disabled Technotherapy Center, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diril E, Menek B, Emir A, Tarakci D, Tarakci E. The Effect of a Video-Based Game Exercise Program on Motor Skills, Proprioception, and Cognitive Functions in Individuals With Intellectual Disabilities. Occup Ther Int. 2025 Jan 30;2025:8410494. doi: 10.1155/oti/8410494. eCollection 2025. PMID 39949506